CLINICAL TRIAL: NCT06557850
Title: Interventional, Open-label, Single-group, Long-term Follow-up Trial of Lu AG22515 in Patients With Moderate-to-severe Thyroid Eye Disease
Brief Title: A Trial Investigating Lu AG22515 in Adult Participants With Moderate-to-Severe Thyroid Eye Disease
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20453A; 2023-508693-29-00 (Other: CTIS)
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Eye Disease
Keywords: Lu AG22515
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lu AG22515 (Experimental): Participants will receive intravenous (IV) administration of Lu AG22515 per a prespecified dosing schedule.
  Interventions: Drug: Lu AG22515

INTERVENTIONS:
Drug: Lu AG22515 — Solution for infusion

SUMMARY:
This trial will evaluate the effects of Lu AG22515 in adult men and women with moderate-to-severe thyroid eye disease (TED). TED is an autoimmune condition closely related to Graves' Disease.

In people with TED, the healthy tissue behind and around the eye becomes inflamed and swollen. One of the key symptoms of TED is proptosis (bulging eyes). The main goal of this trial is to learn whether treatment with Lu AG22515 improves proptosis in participants with moderate-to-severe TED.

ELIGIBILITY:
Inclusion Criteria:

* The participant has Graves' disease associated Thyroid Eye Disease (TED) symptoms characterized by:
* ophthalmologic symptom onset <12 months prior to the Baseline Visit
* proptosis ≥3 millimeter (mm) above normal for race and sex measured using the Hertel exophthalmometer (at the Screening Visit and the Baseline Visit) in the most severe eye
* Clinical Activity Score (CAS) ≥3 in the most severe eye at the Screening Visit.
* The participants must be euthyroid or have mild hypo- or hyperthyroidism (defined as free thyroxin [FT4] and/or free triiodothyronine [FT3] levels not exceeding the normal limits +/-50%) at the Screening Visit.

Exclusion Criteria:

* The participant has a decreased best-corrected visual acuity due to optic neuropathy, defined as a decrease in vision of 2 lines on the Snellen chart, new visual field defect, or colour defect secondary to optic nerve involvement, within 6 months prior to the Screening Visit.
* The participant has corneal decompensation unresponsive to medical management.
* The participant has a decrease in proptosis of ≥2 mm between the Screening Visit and the Baseline Visit.
* The participant has a decrease in CAS of ≥2 points between the Screening Visit and the Baseline Visit.
* The participant has had previous orbital irradiation or surgery for TED.
* The participant requires immediate surgical ophthalmological intervention or has other eye conditions impacting the assessments.
* The participant has contraindications for an magnetic resonance imaging (MRI) scan.
* The participant has an active infection at Baseline or recent serious infection (for example, requiring hospitalization) within 8 weeks prior to the Baseline Visit.
* The participant takes any of the following disallowed or restricted concomitant medications (the list is not comprehensive):
* Disallowed: any investigational products within 30 days or 5 half-lives, whichever is longer, prior to the Screening Visit, systemic corticosteroids within 6 weeks prior to the Screening Visit (topical steroids for dermatological conditions, inhaled or intranasal steroids are allowed), systemic immunosuppressive/immunomodulating drugs (for example, rituximab, tocilizumab, methotrexate, cyclosporine, azathioprine, mycophenolate-sodium/mofetil, Janus kinase inhibitors) within 5 half-lives prior to the Screening Visit, live attenuated vaccines within 30 days prior to the Baseline Visit, biotin within 1 day prior to the Screening Visit.
* Allowed with restriction: stable dose for >3 weeks prior to the Screening Visit of selenium. Inactivated/killed/RNA-based vaccinations are allowed provided they are not administered within 5 days before/after any investigational medicinal product (IMP) trial visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Change in Proptosis from Baseline to Week 24 in the Trial Eye Using the Hertel Exophthalmometer | Baseline, Week 24

SECONDARY OUTCOMES:
Cmax: Maximum Observed Serum Concentration of Lu AG22515 | Predose up to Week 52
Tmax: Time to Maximum Observed Cmax of Lu AG22515 | Predose up to Week 52
Ctrough: Minimum Observed Serum Concentration of Lu AG22515 | Predose up to Week 52
AUC0-infinity: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity of Lu AG22515 | Predose up to Week 52
t½: Apparent Elimination Half-life of Lu AG22515 | Predose up to Week 52
CL: Apparent Total Serum Clearance of Lu AG22515 | Predose up to Week 52
Volume of Distribution of Lu AG22515 | Predose up to Week 52
Number of Participants with Anti-drug Antibodies | Up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — HQ_Medinfo@Lundbeck.com
Locations (6):
- University Clinical Center of The Republic Of Srpska, Banja Luka, Republika Srpska, Bosnia and Herzegovina
- Bulgaria (2):
  - Diagnostic-Consultative Center Alexandrovska, Sofia
  - University Specialized Hospital for Active Treatment in Endocrinology (USHATE) "Acad. Ivan Penchev", Sofia
- Poland (3):
  - Jagiellonian University Medical College, Krakow, Lesser Poland Voivodeship
  - Uniewrsyteckie Centru Kliniczne, Katowice
  - UnivCentrum Zdrowia MDM EB GROUP Sp.zo.o, Warsaw